CLINICAL TRIAL: NCT01550003
Title: A Multicenter, Open-label Study to Assess the Pharmacokinetics, Safety and Efficacy of Certolizumab Pegol in Children and Adolescents With Moderately to Severely Active Polyarticular-course Juvenile Idiopathic Arthritis (JIA)
Brief Title: Pediatric Arthritis Study of Certolizumab Pegol
Acronym: PASCAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB BIOSCIENCES GmbH (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA0043
Expanded Access: NCT03559686 (Available)
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-09

CONDITIONS: Polyarticular-course Juvenile Idiopathic Arthritis (JIA)
Keywords: Cimzia; JIA; Polyarticular; Oligoarticular; Enthesitis-related-Arthritis; Juvenile Idiopathic Arthritis; Juvenile Psoriatic Arthritis; Certolizumab Pegol; PASCAL; CDP870
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Certolizumab Pegol (Experimental): Active treatment with Certolizumab Pegol; dose adjustment is based on weight.
  Interventions: Drug: Certolizumab Pegol (CZP)

INTERVENTIONS:
Drug: Certolizumab Pegol (CZP) — CZP will be administered subcutaneously as a fixed dose based on weight every 2 weeks (Q2W) or every 4 weeks (Q4W) throughout the study.
  CZP will be provided by UCB as a CZP 200 mg/ml solution for single subcutaneous (sc) injection, in a single use prefilled syringe (PFS). Each PFS contains an extractable volume of 0.25 mL, 0.5 mL or 1 mL of CZP solution.
  Eligible subjects will begin with 3 loading doses of CZP followed by a treatment dose for the duration of the study based on the weight range.
  Reduced CZP regimen (after implementation of protocol amendments 4 and 5):
  * 10 to < 20 kg: Loading dose = 50 mg Q2W (1 x 0.25 mL sc); treatment dose = 50 mg Q4W (1 x 0.25 mL sc);
  * 20 to < 40 kg: Loading dose = 100 mg Q2W (1 x 0.5 mL sc,); treatment dose = 50 mg Q2W (1 x 0.25 mL sc);
  * ≥ 40 kg: Loading dose = 200 mg Q2W (1 x 1.0 mL sc); treatment dose = 100 mg Q2W (1 x 0.5 mL sc);
  Other Names: Cimzia
Drug: Certolizumab Pegol (CZP) — CZP will be administered subcutaneously as a fixed dose based on weight every 2 weeks (Q2W) or every 4 weeks (Q4W) throughout the study.
  CZP will be provided by UCB as a CZP 200 mg/ml solution for single subcutaneous (sc) injection, in a single use prefilled syringe (PFS). Each PFS contains an extractable volume of 0.25 mL, 0.5 mL or 1 mL of CZP solution.
  Eligible subjects will begin with 3 loading doses of CZP followed by a treatment dose for the duration of the study based on the weight range.
  Original CZP regimen (prior to implementation of protocol amendments 4 and 5 and after implementation of protocol amendment 9):
  * 10 to < 20 kg: Loading dose = 100 mg Q2W (1 x 0.5 mL sc); treatment dose = 50 mg Q2W (1 x 0.25 mL sc);
  * 20 to < 40 kg: Loading dose = 200 mg Q2W (1 x 1.0 mL sc,); treatment dose = 100 mg Q2W (1 x 0.5 mL sc);
  * ≥ 40 kg: Loading dose = 400 mg Q2W (2 x 1.0 mL sc); treatment dose = 200 mg Q2W (1 x 1.0 mL sc);
  Other Names: Cimzia

SUMMARY:
A Multicenter, Open-label Study to Assess the Pharmacokinetics, Safety and Efficacy of Certolizumab Pegol in Children and Adolescents With Moderately to Severely Active Polyarticular-course Juvenile Idiopathic Arthritis (JIA).

DETAILED DESCRIPTION:
The overall study consists of a Screening Period of up to 4 weeks and an Open-Label Treatment Period which will continue until the approval of the marketing application for the Polyarticular-course Juvenile Idiopathic Arthritis (JIA) indication in the study participant's country or region or until further notice from UCB (approximately 4-6 years duration; depending on region). A Final Visit will be conducted 12 weeks after last dose of study medication. Overall, study visits will occur monthly during the first 6 months and every 2 months afterwards. All patients will receive active treatment with Certolizumab Pegol. The dose will depend on actual weight. Home dosing will be allowed between study visits.

If less than 50 % of the study population achieves an adequate response to the treatment (American College of Rheumatology Pediatric 30 % (PedACR30) response) at Week 16, the study will be entirely discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Study participant is 2 to 17 years of age (inclusive) at Baseline (Visit 2)
* Study participants must weigh ≥10 kg (22lb) at Baseline (Visit 2)
* Study participants must have had onset of signs and symptoms consistent with a diagnosis of Juvenile Idiopathic Arthritis (JIA) (according to the International League of Associations for Rheumatology Classification of Juvenile Idiopathic Arthritis, 2001) and initiation of JIA treatment for at least 6 months prior to Baseline (Visit 2). Eligible JIA categories include: polyarthritis rheumatoid factor-positive, polyarthritis rheumatoid factor-negative, extended oligoarthritis, juvenile psoriatic arthritis, and enthesitis-related arthritis (ERA)
* Study participants must have active polyarticular-course disease, defined as ≥5 joints with active arthritis at Screening and at Baseline
* Study participants must have had an inadequate response to, or intolerance to, at least 1 disease-modifying antirheumatic drug (DMARD) (nonbiologic or biologic). For example, study participant had prior inadequate response to methotrexate (MTX) (based on the Investigator's clinical judgment)
* If the study participant is using MTX, then the study participant must have been on MTX for a minimum of 3 months at Screening. In addition, the dose must have been stable for at least 1 month before Screening at ≥10 to ≤15 mg/m^2 per week. If the study participant is not using MTX, then the treatment must have been previously withdrawn for documented reasons of intolerability or inadequate response
* If the study participant is using oral corticosteroid therapy, the dose must have been stable for at least 7 days prior to the Baseline arthritis assessment at a maximum dose of 10 mg or 0.2 mg/kg prednisone (or equivalent) per day, whichever is the smaller dose

Exclusion Criteria:

* Study participant has previously been exposed to more than 2 biologic agents
* Study participant previously failed to respond to treatment with more than one tumor necrosis factor alpha (TNFα) antagonist drug
* Study participant is currently receiving or has received any experimental (biological or nonbiological) therapy (within or outside a clinical study) in the 3 months or 5 half-lives prior to Baseline (Visit 2), whichever is longer
* Study participant had previous treatment with a biological therapy for juvenile idiopathic arthritis (JIA) that resulted in a severe hypersensitivity reaction or an anaphylactic reaction
* Study participant previously participated in this study or has previously been treated with CZP (whether in a study or not)
* Study participant has a history of systemic JIA, with or without systemic features
* Study participant has a secondary, noninflammatory type of rheumatic disease or of joint pains (eg, fibromyalgia) that in the Investigator's opinion is symptomatic enough to interfere with evaluation of the effect of study medication
* Study participant has other inflammatory arthritis (eg, systemic lupus erythematosus, inflammatory bowel disease-related)
* Study participant has active uveitis or a history of active uveitis within the preceding 6 months
* Study participant has current, chronic or recurrent clinically significant infections
* Study participant has a current sign or symptom which may indicate infection (eg, fever, cough), a history of chronic or recurrent infections within the same organ system (more than 3 episodes requiring antibiotics/antivirals during the 12 months prior to Screening [Visit 1]), had a recent (within the 6 months prior to Screening [Visit 1]) serious or life-threatening infection (including herpes zoster), or is at a high risk of infection in the Investigator's opinion (eg, study participants with leg ulcers, indwelling urinary catheter, and persistent or recurrent chest infections or permanently bed-ridden or wheelchair bound)

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 193 (Actual)
Dates: Start 2012-03-08 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (36):
- United States (20):
  - Ra0043 71, Little Rock, Arkansas
  - Ra0043 79, Los Angeles, California
  - Ra0043 84, San Francisco, California
  - Ra0043 83, Hartford, Connecticut
  - Ra0043 81, Washington D.C., District of Columbia
  - Ra0043 82, Chicago, Illinois
  - Ra0043 90, Chicago, Illinois
  - Ra0043 75, Indianapolis, Indiana
  - Ra0043 80, Hackensack, New Jersey
  - Ra0043 77, Livingston, New Jersey
  - Ra0043 85, New Hyde Park, New York
  - Ra0043 87, New York, New York
  - Ra0043 74, Charlotte, North Carolina
  - Ra0043 76, Durham, North Carolina
  - Ra0043 70, Avon, Ohio
  - Ra0043 73, Cincinnati, Ohio
  - Ra0043 78, Cleveland, Ohio
  - Ra0043 95, Cleveland, Ohio
  - Ra0043 86, Columbus, Ohio
  - Ra0043 89, Portland, Oregon
- RA0043 2, Buenos Aires, Argentina
- Brazil (3):
  - Ra0043 15, Curitiba
  - Ra0043 14, Porto Alegre
  - Ra0043 12, São Paulo
- Canada (3):
  - Ra0043 21, Calgary
  - Ra0043 22, Montreal
  - Ra0043 20, Toronto
- Ra0043 60, Santiago, Chile
- Mexico (4):
  - Ra0043 32, Mexico City
  - Ra0043 31, México
  - Ra0043 30, Monterrey
  - Ra0043 33, San Luis Potosí City
- Russia (4):
  - Ra0043 41, Moscow
  - Ra0043 43, Moscow
  - Ra0043 40, Saint Petersburg
  - Ra0043 42, Tolyatti

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in March 2012 and concluded in April 2024.
Pre-assignment Details: Participant Flow refers to the Safety Set.
Groups:
- Any CZP Dose - Weight Group: 10 - < 20 kg: Participants received Certolizumab Pegol (CZP) subcutaneously (sc) as a fixed dose based on their body weight every 2 weeks (Q2W) or every 4 weeks (Q4W) throughout the study. Participants started with 3 loading doses of CZP at Weeks 0, 2, and 4 followed by a maintenance dose for the duration of the study (maximum up to 12 years).
- Any CZP Dose - Weight Group: 20 - <40 kg; Any CZP Dose - Weight Group: >= 40 kg: Participants received CZP sc as a fixed dose based on their body weight Q2W throughout the study. Participants started with 3 loading doses of CZP at Weeks 0, 2, and 4 followed by a maintenance dose for the duration of the study.
Period: Overall Study
Arm/Group | Any CZP Dose - Weight Group: 10 - < 20 kg | Any CZP Dose - Weight Group: 20 - <40 kg | Any CZP Dose - Weight Group: >= 40 kg
Started | 18 | 63 | 112
Original CZP Dose | 7 | 34 | 64
Reduced CZP Dose | 11 | 29 | 48
Completed | 0 | 0 | 0
Not Completed | 18 | 63 | 112
Not completed — Adverse Event | 0 | 9 | 15
Not completed — Lack of Efficacy | 4 | 11 | 15
Not completed — Protocol Violation | 0 | 3 | 2
Not completed — Lost to Follow-up | 1 | 4 | 8
Not completed — Consent withdrawn | 2 | 11 | 23
Not completed — Missing | 1 | 0 | 2
Not completed — Study closure as announced by sponsor | 7 | 6 | 24
Not completed — Protocol Noncompliance | 1 | 0 | 0
Not completed — Study closure | 0 | 1 | 1
Not completed — Patient reached adulthood | 0 | 1 | 0
Not completed — Early discontinuation at request of sponsor | 0 | 2 | 4
Not completed — Sponsor's order | 0 | 3 | 3
Not completed — Sponsor's decision | 1 | 5 | 4
Not completed — Subject mother passed away | 0 | 1 | 0
Not completed — Discontinuation | 0 | 1 | 0
Not completed — Subject moved to rheumatology and out of study | 0 | 1 | 1
Not completed — Site closure | 0 | 2 | 0
Not completed — Pregnancy | 0 | 1 | 0
Not completed — By medical decision and approved by the sponsor | 0 | 0 | 1
Not completed — Subject is in college/unable to come to visits | 0 | 0 | 1
Not completed — Switching to adult rheumatologist | 0 | 0 | 1
Not completed — Patient transition to adult care | 0 | 0 | 1
Not completed — Subject was able to obtain commercial cimzia | 0 | 0 | 1
Not completed — Treatment or 12 week follow up visit completed | 0 | 0 | 1
Not completed — Per Sponsor request | 1 | 0 | 1
Not completed — Patient not compliance | 0 | 0 | 1
Not completed — Non-compliance | 0 | 0 | 1
Not completed — Study closed | 0 | 1 | 0
Not completed — Transitioned to adult rheumatology | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refers to the Safety Set (SS) which consisted of all study participants in the Enrolled Set (ES) who have received at least 1 dose of study medication.
Groups:
- Any CZP Dose - Weight Group: 10 - <20 kg: Participants received CZP sc as a fixed dose based on their body weight Q2W or Q4W throughout the study. Participants started with 3 loading doses of CZP at Weeks 0, 2, and 4 followed by a maintenance dose for the duration of the study.
- Any CZP Dose - Weight Group: >=40 kg: Participants received CZP sc as a fixed dose based on their body weight Q2W throughout the study. Participants started with 3 loading doses of CZP at Weeks 0, 2, and 4 followed by a maintenance dose for the duration of the study.
- Total: Total of all reporting groups
Arm/Group | Any CZP Dose - Weight Group: 10 - <20 kg | Any CZP Dose - Weight Group: 20 - <40 kg | Any CZP Dose - Weight Group: >=40 kg | Total
Number analyzed (Participants) | 18 | 63 | 112 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.4 (1.3) | 9.1 (2.0) | 14.5 (2.2) | 11.9 (3.8)
Age, Customized [Count of Participants; unit: Participants]
  24 months - <12 years | 18 | 55 | 13 | 86
  12 - <18 years | 0 | 8 | 99 | 107
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 43 | 76 | 130
  Male | 7 | 20 | 36 | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/ Alaska Native | 0 | 1 | 4 | 5
  Asian | 0 | 2 | 3 | 5
  Black or African American | 0 | 0 | 6 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 17 | 53 | 85 | 155
  Other/Mixed | 1 | 7 | 14 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 18 | 27 | 55
  Not Hispanic or Latino | 8 | 45 | 85 | 138

OUTCOME MEASURES:

1. Primary Outcome: Certolizumab Pegol (CZP) Plasma Concentration Level at Week 16
Description: Certolizumab Pegol (CZP) plasma concentration level was measured in micrograms per milliliter (ug/ml).
Time Frame: Week 16
Population: The Pharmacokinetic Per-Protocol (PK-PP) Set was a subset of the SS consisting of those study participants who took at least 1 dose of study medication, provided measurable plasma CZP concentration samples (with recorded sampling date/time or for which date/time can be reasonably assumed). Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: ug/ml
Groups:
- Reduced CZP Dose -Weight Group: 10 - <20 kg: Participants received CZP 50 milligrams (mg) sc Q2W at Weeks 0, 2, and 4 (loading dose) followed by CZP 50 mg sc Q4W (maintenance dose) from Week 8 onwards.
- Reduced CZP Dose - Weight Group: 20 - <40 kg; Original CZP Dose - Weight Group: 10 - <20 kg: Participants received CZP 100 mg sc Q2W at Weeks 0, 2, and 4 (loading dose) followed by CZP 50 mg sc Q2W (maintenance dose) from Week 6 onwards.
- Reduced CZP Dose - Weight Group: >=40 kg; Original CZP Dose - Weight Group: 20 - <40 kg: Participants received CZP 200 mg sc Q2W at Weeks 0, 2, and 4 (loading dose) followed by CZP 100 mg sc Q2W (maintenance dose) from Week 6 onwards.
- Original CZP Dose - Weight Group: >=40 kg: Participants received CZP 400 mg sc Q2W at Weeks 0, 2, and 4 (loading dose) followed by CZP 200 mg sc Q2W (maintenance dose) from Week 6 onwards.
Arm/Group | Reduced CZP Dose -Weight Group: 10 - <20 kg | Reduced CZP Dose - Weight Group: 20 - <40 kg | Reduced CZP Dose - Weight Group: >=40 kg | Original CZP Dose - Weight Group: 10 - <20 kg | Original CZP Dose - Weight Group: 20 - <40 kg | Original CZP Dose - Weight Group: >=40 kg
Number analyzed (Participants) | 10 | 24 | 36 | 5 | 29 | 49
ug/ml | 1.6166 [0.4720 to 5.5368] | 9.2277 [5.1453 to 16.5491] | 13.8928 [11.0030 to 17.5416] | 22.9060 [13.3380 to 39.3374] | 25.7752 [16.9024 to 39.3058] | 33.5680 [25.7883 to 43.6945]

2. Primary Outcome: Certolizumab Pegol (CZP) Plasma Concentration Level at Week 48
Description: Certolizumab Pegol (CZP) plasma concentration level was measured in ug/mL.
Time Frame: Week 48
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ug/ml
Arm/Group | Reduced CZP Dose -Weight Group: 10 - <20 kg | Reduced CZP Dose - Weight Group: 20 - <40 kg | Reduced CZP Dose - Weight Group: >=40 kg | Original CZP Dose - Weight Group: 10 - <20 kg | Original CZP Dose - Weight Group: 20 - <40 kg | Original CZP Dose - Weight Group: >=40 kg
Number analyzed (Participants) | 9 | 24 | 31 | 2 | 12 | 25
ug/ml | 4.7404 [1.7596 to 12.7710] | 8.4459 [5.0002 to 14.2661] | 12.2987 [8.6950 to 17.3962] | NA [NA to NA] — As pre-specified in the SAP, Geometric Mean and 95% confidence interval (CI) were not calculated if less than 3 concentration were available or if the below the lower limit of quantification (LLOQ) was greater than (>) 1/3. | 20.7048 [11.1744 to 38.3636] | 25.5940 [14.6913 to 44.5878]

3. Primary Outcome: Number of Participants With Anti-Certolizumab Pegol (Anti-CZP) Antibody Level at Week 16
Description: Number of participants with anti-CZP antibodies were reported.
Time Frame: Week 16
Population: Safety Set (SS) consisted of all study participants in the Enrolled Set (ES) who have received at least 1 dose of study medication. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Reduced CZP Dose: Participants received reduced CZP sc as a fixed dose based on their body weight Q2W or Q4W throughout the study. Participants started with 3 loading doses of CZP at Weeks 0, 2, and 4 followed by a maintenance dose for the duration of the study.
- Original CZP Dose: Participants received original CZP sc as a fixed dose based on their body weight Q2W throughout the study. Participants started with 3 loading doses of CZP at Weeks 0, 2, and 4 followed by a maintenance dose for the duration of the study.
Arm/Group | Reduced CZP Dose | Original CZP Dose
Number analyzed (Participants) | 84 | 97
Participants | 69 | 77

4. Primary Outcome: Number of Participants With Anti-Certolizumab Pegol (Anti-CZP) Antibody Level at Week 48
Description: Number of participants with anti-CZP antibodies were reported.
Time Frame: Week 48
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced CZP Dose | Original CZP Dose
Number analyzed (Participants) | 72 | 60
Participants | 58 | 47

5. Primary Outcome: Number of Participants With Serious Treatment-emergent Adverse Events (TEAEs) During the Study
Description: A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose: results in deaths, is life-threatening, requires in patient hospitalization or prolongation of existing hospitalization, is a congenital anomaly or birth defect and other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above. TEAEs are defined as AEs starting on or after first administration of CZP and up to 70 days after last dose of study medication.
Time Frame: From Baseline (Week 0) up to the Final Visit (70 days after final dose of CZP) (maximum up to 12 years)
Population: Safety Set (SS) consisted of all study participants in the Enrolled Set (ES) who have received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Any CZP Dose - Weight Group: 10 - <20 kg | Any CZP Dose - Weight Group: 20 - <40 kg | Any CZP Dose - Weight Group: >=40 kg
Number analyzed (Participants) | 18 | 63 | 112
Participants | 5 | 20 | 21

6. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Leading to Permanent Withdrawal of the Investigational Medicinal Product (IMP) During the Study
Description: An AE is any untoward medical occurrence in a patient or clinical investigation study participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an IMP, whether or not related to the IMP. TEAEs are defined as AEs starting on or after first administration of CZP and up to 70 days after last dose of study medication. TEAEs leading to permanent withdrawal of the IMP during the study were reported in this outcome measure.
Time Frame: From Baseline (Week 0) up to the Final Visit (70 days after final dose of CZP) (maximum up to 12 years)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Any CZP Dose - Weight Group: 10 - <20 kg | Any CZP Dose - Weight Group: 20 - <40 kg | Any CZP Dose - Weight Group: >=40 kg
Number analyzed (Participants) | 18 | 63 | 112
Participants | 0 | 9 | 16

7. Secondary Outcome: Percentage of Participants Meeting American College of Rheumatology Pediatric 30 % (PedACR30) Response Criteria at Week 16
Description: PedACR30-at least 30% improvement from baseline in 3 of any 6 core set measures, with no more than 1 of remaining variables worsening by >30%:
  * Number of joints with active arthritis
  * Number of joints with limitation of range of motion
  * Physician's Global Assessment of Disease Activity (using visual analog scale (VAS): 100mm; 0= very good, and 100= very poor)
  * CHAQ (30 questions, 8 domains, scores for each domain are averaged to calculate total score [ 0= no disability to 3= very severe disability])
  * Parent's Global Assessment of Overall Well-Being (using VAS: 100mm; 0= Very well to 100= Very poor)
  * C-reactive protein (CRP)
Time Frame: Week 16
Population: Full analysis set (FAS): all study participants in SS who have no more than one of 6 core components missing at baseline (count of joints with active arthritis, count of joints with limitation of range of motion, Physician's Global Assessment of Disease Activity score, CHAQ score, Parent's Global Assessment of Overall Well-Being score and CRP result) for calculating PedACR30/50/70/90.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Any CZP Dose - Weight Group: 10 - <20 kg | Any CZP Dose - Weight Group: 20 - <40 kg | Any CZP Dose - Weight Group: >=40 kg
Number analyzed (Participants) | 18 | 63 | 112
percentage of participants | 83.3 [58.6 to 96.4] | 77.8 [65.5 to 87.3] | 79.5 [70.8 to 86.5]

8. Secondary Outcome: Percentage of Participants Meeting American College of Rheumatology Pediatric 50 % (PedACR50) Response Criteria at Week 16
Description: PedACR50- at least 50% improvement from baseline in 3 of any 6 core set measures, with no more than 1 of remaining variables worsening by >30%:
  * Number of joints with active arthritis
  * Number of joints with limitation of range of motion
  * Physician's Global Assessment (PGA) of Disease Activity (using VAS: 100mm; 0= very good, and 100= very poor)
  * Childhood Health Assessment Questionnaire (CHAQ) (30 questions, 8 domains, scores for each domain are averaged to calculate total score [ 0= no disability to 3= very severe disability])
  * Parent's Global Assessment of Overall Well-Being (using VAS: 100mm; 0= Very well to 100= Very poor)
  * CRP
Time Frame: Week 16
Population: FAS:all study participants in SS who have no more than one of 6 core components missing at baseline (count of joints with active arthritis, count of joints with limitation of range of motion, PGA of Disease Activity score, CHAQ score, Parent's Global Assessment of Overall Well-Being score and CRP result) for calculating PedACR30/50/70/90.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Any CZP Dose - Weight Group: 10 - <20 kg | Any CZP Dose - Weight Group: 20 - <40 kg | Any CZP Dose - Weight Group: >=40 kg
Number analyzed (Participants) | 18 | 63 | 112
percentage of participants | 66.7 [41.0 to 86.7] | 71.4 [58.7 to 82.1] | 74.1 [65.0 to 81.9]

9. Secondary Outcome: Percentage of Participants Meeting American College of Rheumatology Pediatric 70 % (PedACR70) Response Criteria at Week 16
Description: PedACR70- at least 70% improvement from baseline in 3 of any 6 following core set measures, with no more than 1 of remaining variables worsening by >30%:
  * Number of joints with active arthritis
  * Number of joints with limitation of range of motion
  * Physician's Global Assessment of Disease Activity (using VAS: 100mm; 0= very good, and 100= very poor)
  * CHAQ (30 questions, 8 domains, scores for each domain are averaged to calculate total score [ 0= no disability to 3= very severe disability])
  * Parent's Global Assessment of Overall Well-Being (using VAS: 100mm; 0= Very well to 100= Very poor)
  * CRP
Time Frame: Week 16
Population: FAS consisted of all study participants in SS who have no more than one of 6 core components missing at baseline (count of joints with active arthritis, count of joints with limitation of range of motion, Physician's Global Assessment of Disease Activity score, CHAQ score, Parent's Global Assessment of Overall Well-Being score and CRP result) for calculating PedACR30/50/70/90.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Any CZP Dose - Weight Group: 10 - <20 kg | Any CZP Dose - Weight Group: 20 - <40 kg | Any CZP Dose - Weight Group: >=40 kg
Number analyzed (Participants) | 18 | 63 | 112
percentage of participants | 44.4 [21.5 to 69.2] | 57.1 [44.0 to 69.5] | 54.5 [44.8 to 63.9]

10. Secondary Outcome: Percentage of Participants Meeting American College of Rheumatology Pediatric 90 % (PedACR90) Response Criteria at Week 16
Description: PedACR90- at least 90% improvement from baseline in 3 of any 6 following core set measures, with no more than 1 of remaining variables worsening by >30%:
  * Number of joints with active arthritis
  * Number of joints with limitation of range of motion
  * Physician's Global Assessment of Disease Activity (using VAS: 100mm; 0= very good, and 100= very poor)
  * CHAQ (30 questions, 8 domains, scores for each domain are averaged to calculate total score [ 0= no disability to 3= very severe disability])
  * Parent's Global Assessment of Overall Well-Being (using VAS: 100mm; 0= Very well to 100= Very poor)
  * CRP
Time Frame: Week 16
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Any CZP Dose - Weight Group: 10 - <20 kg | Any CZP Dose - Weight Group: 20 - <40 kg | Any CZP Dose - Weight Group: >=40 kg
Number analyzed (Participants) | 18 | 63 | 112
percentage of participants | 22.2 [6.4 to 47.6] | 25.4 [15.3 to 37.9] | 29.5 [21.2 to 38.8]

ADVERSE EVENTS:
Time Frame: From Baseline (Week 0) up to the Final Visit (70 days after final dose of CZP) (maximum up to 12 years)
Description: TEAEs were defined as AEs starting on or after first administration of CZP and up to 70 days after last dose of study medication. Safety Set (SS) consisted of all study participants in the Enrolled Set (ES) who have received at least 1 dose of study medication.
Arm/Group | Any CZP Dose - Weight Group: 10 - <20 kg | Any CZP Dose - Weight Group: 20 - <40 kg | Any CZP Dose - Weight Group: >=40 kg
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/63 | 3/112
Serious Adverse Events (participants affected / at risk) | 5/18 | 20/63 | 21/112
Other Adverse Events (participants affected / at risk) | 16/18 | 59/63 | 98/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Any CZP Dose - Weight Group: 10 - <20 kg (N=18) | Any CZP Dose - Weight Group: 20 - <40 kg (N=63) | Any CZP Dose - Weight Group: >=40 kg (N=112)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Adrenal suppression (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 5 (5) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Serratia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tuberculosis liver (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Varicella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hair follicle tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Idiopathic generalised epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pregnancy on contraceptive (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Drug abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Any CZP Dose - Weight Group: 10 - <20 kg (N=18) | Any CZP Dose - Weight Group: 20 - <40 kg (N=63) | Any CZP Dose - Weight Group: >=40 kg (N=112)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 5 (6) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 4 (5) | 3 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Lichen spinulosus (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 3 (5) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 1 (1) | 1 (2)
Uveitis (Eye disorders) | 1 (1) | 2 (3) | 0 (0)
Iritis (Eye disorders) | 1 (2) | 0 (0) | 1 (2)
Hypermetropia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 6 (8) | 14 (22)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 5 (5) | 13 (14)
Nausea (Gastrointestinal disorders) | 1 (2) | 3 (5) | 13 (19)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 8 (9) | 8 (12)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (2) | 4 (4)
Dental caries (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Retained deciduous tooth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Salivary gland mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (6) | 12 (18) | 11 (20)
Injection site pain (General disorders) | 2 (2) | 5 (25) | 10 (30)
Fatigue (General disorders) | 0 (0) | 5 (6) | 9 (11)
Injection site reaction (General disorders) | 0 (0) | 1 (2) | 6 (9)
Condition aggravated (General disorders) | 1 (1) | 1 (1) | 2 (2)
Cyst (General disorders) | 1 (1) | 0 (0) | 2 (2)
Drug intolerance (General disorders) | 1 (1) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 4 (8) | 17 (46) | 32 (68)
Upper respiratory tract infection (Infections and infestations) | 4 (11) | 16 (41) | 28 (62)
Respiratory tract infection (Infections and infestations) | 1 (6) | 12 (22) | 11 (15)
Viral infection (Infections and infestations) | 2 (2) | 7 (12) | 13 (17)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 10 (16) | 9 (18)
Pharyngitis (Infections and infestations) | 1 (1) | 9 (11) | 7 (9)
Sinusitis (Infections and infestations) | 0 (0) | 5 (6) | 12 (20)
Tonsillitis (Infections and infestations) | 2 (3) | 9 (9) | 6 (11)
Influenza (Infections and infestations) | 1 (1) | 5 (8) | 10 (16)
Gastroenteritis (Infections and infestations) | 0 (0) | 4 (4) | 11 (19)
Rhinitis (Infections and infestations) | 0 (0) | 8 (12) | 7 (9)
Urinary tract infection (Infections and infestations) | 0 (0) | 4 (4) | 10 (23)
Bronchitis (Infections and infestations) | 1 (1) | 6 (6) | 6 (6)
Conjunctivitis (Infections and infestations) | 2 (2) | 3 (3) | 7 (7)
Latent tuberculosis (Infections and infestations) | 2 (2) | 7 (7) | 2 (2)
Ear infection (Infections and infestations) | 2 (2) | 4 (5) | 4 (6)
Varicella (Infections and infestations) | 4 (4) | 4 (4) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 6 (9)
Respiratory tract infection viral (Infections and infestations) | 2 (2) | 4 (4) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)
Impetigo (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)
Viral pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 4 (5)
Otitis media acute (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Bacteriuria (Infections and infestations) | 1 (1) | 1 (2) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (3) | 0 (0)
Viral rash (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
Ascariasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 5 (6) | 9 (11)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (4) | 6 (7)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 3 (3)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 2 (5)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 5 (8) | 10 (12)
Alanine aminotransferase increased (Investigations) | 1 (1) | 5 (5) | 9 (12)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 6 (8)
C-reactive protein increased (Investigations) | 2 (2) | 1 (2) | 6 (6)
Hepatic enzyme increased (Investigations) | 2 (2) | 1 (1) | 6 (7)
Mycobacterium tuberculosis complex test positive (Investigations) | 1 (1) | 2 (2) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 12 (19) | 20 (37)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (11) | 10 (17)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (6) | 10 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 6 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 5 (5)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (6)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 7 (16) | 30 (56)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 6 (9)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 8 (11)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 7 (7)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 1 (3) | 3 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 10 (16) | 11 (21)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (12) | 15 (19)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (8) | 6 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 7 (18)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (4) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (7) | 10 (13)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (7) | 2 (2)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/03/NCT01550003/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/03/NCT01550003/SAP_001.pdf